CLINICAL TRIAL: NCT04701892
Title: Central Sensitisation in Post Covid-19 Infection Patients: a Prospective Cohort Study
Brief Title: poSt Covid-19 Infection centraL Sensitisation 2
Acronym: SILENT 2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: SILENT 2
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 infected patients: In this study male and female patients who were previously infected with covid-19 will be included. Patients will only be eligible if they had a positive covid-19 test before inclusion in the study. More specifically, only patients who had a positive COVID-19 test 2 to 8 weeks before study inclusion are eligible.
  Interventions: Other: Indicators of central sensitisation

INTERVENTIONS:
Other: Indicators of central sensitisation — Indicators of central sensitisation, assessed by the Central Sensitization Inventory

SUMMARY:
The aim of this study is to evaluate whether there are indicators of central sensitisation in patients post covid-19 infection.

DETAILED DESCRIPTION:
The COVID-19 pandemic is currently a serious global public health concern. This disease is caused by a novel coronavirus which was first discovered in Wuhan, China in 2019 and later spread rapidly throughout the world. Symptoms of the disease can manifest as fever, cough, encephalitis, myalgia, fatigue, muscle weakness, arthralgia, anosmia, and impairment in other bodily functions in the acute phase. In 17% to 67% of cases, COVID-19 patients will develop acute respiratory distress syndrome (ARDS) and critical illness. Besides the impact on the respiratory system, coronaviruses have an effect on other systems including the central nervous system, cardiovascular system, musculoskeletal system, and gastrointestinal system.

The term central sensitivity syndrome (CSS) describes a group of medically nonspecific disorders, such as fibromyalgia, chronic fatigue syndrome, and irritable bowel syndrome, for which central sensitivity might be a common etiology. Despite the lack of a solid outcome measurement, the Central Sensitization Inventory (CSI) was previously introduced as a screening instrument for clinicians to help identify patients with a CSS. Furthermore, quantitative sensory testing can be used to identify and quantify sensory disfunctions by evaluating a variety of parameters including pain thresholds, temporal summation, and conditioned pain modulation (CPM). Previous research in patients with chronic pain resulted in less efficacious CPM, increased nociceptive facilitation and decreased pain thresholds.

In post covid-19 patients, potential long-term secondary effects on the musculoskeletal system such as muscle weakness, decreased muscle mass, and myopathies have been brought under attention. Persisting symptoms are a frequently reported complaint in patients recovered from COVID-19 infection with at least 1 symptom, particularly fatigue and dyspnea. Fatigue is also one of the core symptoms in central sensitisation disorders, leading to the hypothesis that central sensitisation might be the underlying common etiology in chronic pain patients and patients post COVID-19 infection. Therefore, the aim of this study is to evaluate whether there are indicators of central sensitisation in patients post covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosed covid-19 infection that took place 2-8 weeks before study inclusion.
* Cognitive and language functioning enabling coherent communication between the researcher and the participant.
* French-or Dutch speaking persons.

Exclusion Criteria:

* Covid-19 infection > 8 weeks ago.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients who were previously infected with covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms of Central Sensitisation | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Symptoms of central sensitisation will be measured with the Central Sensitization Inventory.

SECONDARY OUTCOMES:
Pressure pain thresholds | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Pressure pain thresholds will be measured at the trapezius and rectus femoris muscles with an algometer.
Temporal summation | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Temporal summation will be measured with 10 consecutive pressure pulses at the trapezius and rectus femoris muscles with an algometer.
Descending nociceptive inhibition | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Descending nociceptive inhibition will be measured with a conditioned pain modulation protocol with algometer as test stimulus and the cold pressor task.
Functionality and disability | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Functional status will be evaluated by the Post-COVID-19 Functional Status Scale.
Functionality and disability | The change between baseline, 3 months, 6 months (primary time endpoint) and 12 months
  Level of dyspnea during activities of daily living will be evaluated by the London chest Activity of Daily Living scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium